CLINICAL TRIAL: NCT00000639
Title: A Randomized Double Blind Protocol Comparing Amphotericin B With Flucytosine to Amphotericin B Alone Followed by a Comparison of Fluconazole and Itraconazole in the Treatment of Acute Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 159; FDA 235A; MSG Study 17; 11134 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Drug Evaluation; Drug Therapy, Combination; Fluconazole; Flucytosine; Acquired Immunodeficiency Syndrome; Amphotericin B; Brain Diseases
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome; Brain Diseases | interventions — Itraconazole; Flucytosine; Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Itraconazole
Drug: Flucytosine
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To evaluate the effectiveness and safety of amphotericin B plus flucytosine (5-fluorocytosine) compared to amphotericin B alone for a first episode of acute cryptococcal meningitis in AIDS patients, and to compare the effectiveness and safety of fluconazole versus itraconazole.

At least 10 percent of patients with a low CD4 count and HIV infection will develop meningitis due to Cryptococcus neoformans. More effective treatments than the standard therapy need to be explored.

DETAILED DESCRIPTION:
At least 10 percent of patients with a low CD4 count and HIV infection will develop meningitis due to Cryptococcus neoformans. More effective treatments than the standard therapy need to be explored.

Patients are selected by a randomization process to take amphotericin B intravenously (in the vein), for 14 days, and either placebo (ineffective substance) or flucytosine for 14 days. Then patients are again selected by a randomization process to take either (1) fluconazole for a total of 8 weeks plus itraconazole placebo; or (2) itraconazole for a total of 8 weeks plus fluconazole placebo.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Interruption of myelosuppressive therapies and/or administration of erythropoietin, at discretion of investigator, to maintain hemoglobin = or > 7 g/dl.
* Adjunctive corticosteroids may be administered during the triazole phase for patients who develop Pneumocystis carinii pneumonia and meet the prescribed criteria.
* Hydrocortisone, not to exceed 50 mg/day, during the amphotericin phase.
* Aerosolized pentamidine or systemic chemoprophylaxis for Pneumocystis carinii pneumonia should be given to all patients with a CD4 count < 200 cells/mm3.
* Antiretroviral drugs (including zidovudine (AZT), didanosine (ddI), dideoxycytidine (ddC)) after patient has tolerated oral triazole for one week (after 3 weeks of study treatment).
* Maintenance treatment (except for rifamycins) for other opportunistic infections such as cytomegalovirus (CMV) retinitis, cerebral toxoplasmosis or mycobacterial infections, provided that their hematologic and hepatic values are stable and they meet the entry criteria.

Concurrent Treatment:

Allowed:

- Transfusion, at discretion of investigator, to maintain hemoglobin = or > 7 g/dl.

Patients must have:

* HIV infection.
* Primary episode of acute cryptococcal meningitis.
* Willing to participate in the study for a full 10 weeks and either be able to give informed consent or have a family member or guardian able to give informed consent.

Prior Medication:

Allowed:

Fluconazole prophylaxis, not exceeding 200 mg/day.

Risk Behavior:

Allowed:

- History of high-risk behavior for HIV infection (bisexual or homosexual men, intravenous drug abusers) and their sexual partners.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Inability to take oral medication (if necessary, flucytosine and flucytosine placebo may be administered via nasogastric tube during the amphotericin phase).
* History of hypersensitivity to imidazole or triazole compounds.
* Active hepatitis (viral, drug-induced, or other) defined by progressive worsening of hepatic enzymes to grade 3 or 4 toxicity on at least two occasions.
* Comatose.
* Concurrent CNS disease which, in the opinion of the investigator, would interfere with assessment of response.

Concurrent Medication:

Excluded:

* Continued treatment with H2 blockers (ranitidine (Zantac), cimetidine (Tagamet), omeprazole (Prilosec), nizatidine (Axid), famotidine (Pepcid)).
* Antacids and didanosine (ddI) within 2 hours of triazole administration.
* Rifampin, rifabutin (Ansamycin), and other rifamycin derivatives, phenytoin (Dilantin), phenobarbital, or carbamazepine (Tegretol).
* Other systemic antifungal agents.

Prior Medication:

Excluded:

* Amphotericin, > 1 mg/kg, or fluconazole or ketoconazole, > 1200 mg, as prior treatment for current primary episode of acute cryptococcal meningitis or treatment started for this episode more than 72 hours prior to enrollment into study.
* Phenytoin (Dilantin), carbamazepine (Tegretol), phenobarbital, rifabutin (Ansamycin), rifampin or other rifamycins within the last 15 days.

Patients may not have:

* Inability to take oral medication (if necessary, flucytosine and flucytosine placebo may be administered via nasogastric tube during the amphotericin phase).
* History of hypersensitivity to imidazole or triazole compounds.
* Active hepatitis.
* Patients who are comatose.
* Concurrent CNS disease which, in the opinion of the investigator, would interfere with assessment of response.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1997-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: van der Horst C, Study Chair; Saag M, Study Chair
Locations (24):
- United States (24):
  - USC CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] van der Horst CM, Saag MS, Cloud GA, Hamill RJ, Graybill JR, Sobel JD, Johnson PC, Tuazon CU, Kerkering T, Moskovitz BL, Powderly WG, Dismukes WE. Treatment of cryptococcal meningitis associated with the acquired immunodeficiency syndrome. National Institute of Allergy and Infectious Diseases Mycoses Study Group and AIDS Clinical Trials Group. N Engl J Med. 1997 Jul 3;337(1):15-21. doi: 10.1056/NEJM199707033370103. PMID 9203426
- [Background] Powderly WG. Recent advances in the management of cryptococcal meningitis in patients with AIDS. Clin Infect Dis. 1996 May;22 Suppl 2:S119-23. doi: 10.1093/clinids/22.supplement_2.s119. PMID 8722838
- [Background] Powderly WG, Tuazon C, Cloud GA, Saag MS, Van Der Horst C. Serum and CSF cryptococcal antigen in management of cryptococcal meningitis in AIDS. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:66 (abstract no 6)